CLINICAL TRIAL: NCT06800105
Title: Dysregulation of Whole-body Metabolism in Ovarian Cancer: A Longitudinal Study
Status: Recruiting | Type: Observational
Sponsor: University of Tennessee Graduate School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 5023
Record Dates: First submitted 2023-10-30; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Ovary Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with presumed ovarian cancer: Patients with presumed ovarian cancer will complete three, 4-hour study visits at the following time points:
  * The 1st visit will occur before treatment.
  * The 2nd visit will occur after about half of the planned treatment as been completed.
  * The 3rd visit will occur 4-8 weeks after the completion of treatment.
  Interventions: Other: High fat smoothie

INTERVENTIONS:
Other: High fat smoothie — Participants will consume a standardized 490 kcal high-fat smoothie, consisting of 57% fat, 23% carbohydrate, and 20% protein.

SUMMARY:
Minimal information is available regarding changes in whole-body metabolism in ovarian cancer patients, and no study has assessed whole-body lipid metabolism in this patient population. In this pilot study we will assess fasting and postprandial lipid metabolism of ovarian cancer patients before, during, and after treatment via indirect calorimetry.

DETAILED DESCRIPTION:
Ovarian cancer is one of the deadliest gynecological diseases, with a 5-year survival rate of only 49%. It is well established that cancer cells have fundamentally altered metabolism, which contributes to proliferation and metastasis. Recent findings in the field have recognized that lipid metabolism is altered in ovarian cancer cells, with cells utilizing lipids as a primary energy source. Due to the high demand of energy from tumor cells, it's possible that other non-malignant tissues could reprogram their metabolism to create an environment that supports tumor growth. Minimal information is available regarding changes in whole-body metabolism in ovarian cancer patients, and no study has assessed whole-body lipid metabolism in this patient population. In this pilot study we will assess fasting and postprandial lipid metabolism of ovarian cancer patients before, during, and after treatment via indirect calorimetry. Markers of metabolism (e.g. glucose, blood lipids, lactate) will be assessed at each timepoint. This is a clinically significant project as understanding the full scope of dysregulated lipid metabolism in ovarian cancer patients will allow the identification of potential targets for treatment. The primary purpose is to assess feasibility and acceptability of this study protocol designed to collect pilot data and assess the metabolic profile and lipid metabolism of patients with presumed ovarian cancer. The secondary purpose of this project is to collect pilot data and assess the metabolic profile and lipid metabolism of patients with presumed ovarian cancer. A tertiary goal of this project is to collect additional pilot data to better understand the potential link between metabolic health and other factors related to metabolic health among patients with ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age >18
* Presumed ovarian cancer diagnosis (i.e. those being clinically evaluated for suspicion of ovary cancer)
* Planned treatment course for ovarian cancer involving cytoreductive surgery followed by chemotherapy
* Availability to commit to attending all study visits
* Internet access and consistent access to phone/email/text communication

Exclusion Criteria:

* Pregnancy
* Inability to provide voluntary informed consent
* Inability to consume the pre-study visit meal/snack and/or the study visit meal due to strict dietary restrictions
* Illicit substance use (e.g. cocaine, methamphetamines, heroin, street drugs) - marijuana and CBD oil and related supplements will be considered on a case-by-case basis by the principal investigators
* Circumstances and/or medical condition that would limit compliance with study requirements and protocol, as determined by the principal investigators

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Being clinically treated for gynecologic malignancy
Study Population: Patients being treated clinically for gynecologic malignancy
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility assessed by attrition | 60 months
  Feasibility assessed by ≤20% attrition (yes/no), defined as the percentage of enrolled participants, that are able to complete all three study visits.
Feasibility and acceptability assessed by protocol adherence | 60 months
  Feasibility and acceptability assessed by ≥75% protocol adherence (yes/no) specifically measured by:
  Ability of the participant to consume pre-study visit meal Ability of the participant to consume study visit smoothie in 5 minutes Ability of the participant to complete the 4 metabolic assessments during the study visit Ability of the participant to complete surveys during the study visit Ability of the participant to arrive on time and leave at the planned time for the study visit Ability of the study team to coordinate delivery of the pre-study visit meal to participant

SECONDARY OUTCOMES:
Fasting resting energy expenditure | Immediately at the beginning of the study visit
  Fasting resting energy expenditure (Kcal/D) assessed using indirect calorimetry.
Fasting respiratory quotient (RQ) | Immediately at the beginning of the study visit
  Fasting respiratory quotient (RQ) assessed using indirect calorimetry
Fasting carbon dioxide production | Immediately at the beginning of the study visit
  Fasting carbon dioxide production (VCO2) (ml/min) assessed using indirect calorimetry.
Fasting oxygen consumption | Immediately at the beginning of the study visit
  Fasting oxygen consumption (VO2)(ml/min) assessed using indirect calorimetry.
Fasting capillary blood glucose | Immediately at the beginning of the study visit
  Fasting capillary blood glucose (mg/dL)
Fasting capillary blood lactate | Immediately at the beginning of the study visit
  Fasting capillary blood lactate (mmol/L)
1 hour resting energy expenditure | Assessed at 1 hour post- high-fat smoothie consumption
  1 hour resting energy expenditure (Kcal/D) assessed using indirect calorimetry.
1 hour respiratory quotient (RQ) | Assessed at 1 hour post- high-fat smoothie consumption
  1 hour respiratory quotient (RQ) assessed using indirect calorimetry
1 hour carbon dioxide production | Assessed at 1 hour post- high-fat smoothie consumption
  1 hour carbon dioxide production (VCO2) (ml/min) assessed using indirect calorimetry.
1 hour oxygen consumption | Assessed at 1 hour post- high-fat smoothie consumption
  1 hour oxygen consumption (VO2)(ml/min) assessed using indirect calorimetry.
1 hour capillary blood glucose | Assessed at 1 hour post- high-fat smoothie consumption
  1 hour capillary blood glucose (mg/dL)
1 hour capillary blood lactate | Assessed at 1 hour post- high-fat smoothie consumption
  1 hour capillary blood lactate (mmol/L)
2 hour resting energy expenditure | Assessed at 2 hours post- high-fat smoothie consumption
  2 hour resting energy expenditure (Kcal/D) assessed using indirect calorimetry.
2 hour respiratory quotient (RQ) | Assessed at 2 hour post- high-fat smoothie consumption
  2 hour respiratory quotient (RQ) assessed using indirect calorimetry
2 hour carbon dioxide production | Assessed at 2 hours post- high-fat smoothie consumption
  2 hour carbon dioxide production (VCO2) (ml/min) assessed using indirect calorimetry.
2 hour oxygen consumption | Assessed at 2 hours post- high-fat smoothie consumption
  2 hour oxygen consumption (VO2)(ml/min) assessed using indirect calorimetry.
2 hour capillary blood glucose | Assessed at 2 hours post- high-fat smoothie consumption
  2 hour capillary blood glucose (mg/dL)
2 hour capillary blood lactate | Assessed at 2 hours post- high-fat smoothie consumption
  2 hour capillary blood lactate (mmol/L)
3 hour resting energy expenditure | Assessed at 3 hours post- high-fat smoothie consumption
  3 hour resting energy expenditure (Kcal/D) assessed using indirect calorimetry.
3 hour respiratory quotient (RQ) | Assessed at 3 hours post- high-fat smoothie consumption
  3 hour respiratory quotient (RQ) assessed using indirect calorimetry
3 hour carbon dioxide production | Assessed at 3 hours post- high-fat smoothie consumption
  3 hour carbon dioxide production (VCO2) (ml/min) assessed using indirect calorimetry.
3 hour oxygen consumption | Assessed at 3 hours post- high-fat smoothie consumption
  3 hour oxygen consumption (VO2)(ml/min) assessed using indirect calorimetry.
3 hour capillary blood glucose | Assessed at 3 hours post- high-fat smoothie consumption
  3 hour capillary blood glucose (mg/dL)
3 hour capillary blood lactate | Assessed at 3 hours post- high-fat smoothie consumption
  3 hour capillary blood lactate (mmol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee Graduate School of Medicine, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided
Datasets will not be publicly available but can be shared by request.